CLINICAL TRIAL: NCT00793052
Title: Etodalac, Etoricoxib and Dexamethasone for Prevention of Pain ,Swelling and Trismus Following Third Molar Surgery: A Prospective, Double-Blind Study
Brief Title: Etodalac, Etoricoxib and Dexamethasone for Prevention of Pain ,Swelling and Trismus Following Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Oral and maxillofacial surgery unit, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-08-BS-062-CTIL
Record Dates: First submitted 2008-10-29; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Trismus; Edema; Pain
Keywords: trismus; Edema; pain
MeSH Terms: conditions — Trismus; Edema; Pain | interventions — Etoricoxib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Etodalac, Etoricoxib and Dexamethasone

INTERVENTIONS:
Drug: Etodalac, Etoricoxib and Dexamethasone — Dexamethasone sodium phosphate 8 mg 1 hour before the extraction, 4 mg the day after the extraction and another 4 mg at second day to the extraction.
  Etoricoxib 120 mg 1 hour before the extraction, 120 mg the day after the extraction and another 120 mg at second day to the extraction.
  Etodalac 600 mg 1 hour before the extraction, 600 mg the day after the extraction and another 600 mg at second day to the extraction.

SUMMARY:
The purpose of this study is to determine whether Etodalac, Etoricoxib and Dexamethasone are effective for Prevention of Pain ,Swelling and Trismus Following Third Molar Surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients who are refered for third molar extraction to our center
* Must be able to swallow tablets

Exclusion Criteria:

* Diabetes mellitus
* Thyroid diseases
* Cardiovascular diseases
* renal diseases
* hepatic diseases
* respiratory system diseases
* adrenal diseases
* Allergy to Etodalac, Etoricoxib or Dexamethasone
* Gastric ulcers
* psychiatric diseases
* Pregnant or breast feeding womans

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
PAIN- By VAS graded from 1-10 TRISMUS- By MAX mouth opening from the first incisors adages POST OPERATIVE SWELLing - By measurement the distance between the Right and LEFT ear's tragus | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: benjamin Shlomi, DMD, Study Chair — MAXILLOFACIAL SURGERY - TASMC